CLINICAL TRIAL: NCT03670433
Title: Medication Reconciliation for Patients Over 65 Years Old : Cost Analysis of the Process Implemented in the Polyvalent Internal Medical Unit of Rennes University Hospital
Acronym: CONTEMPS
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_3081
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Medication Reconciliation
Keywords: Medication reconciliation; Care path; Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted in the Polyvalent Internal Medical Unit: Patients over 65 years old admitted in the Polyvalent Internal Medical Unit (UMIP) of Rennes University Hospital between 09/04/2017 and 10/31/2017 or going back home or to a rehabilitation service during the same period.
  Cost analysis of medication reconciliation.
  Interventions: Other: Cost analysis of medication reconciliation

INTERVENTIONS:
Other: Cost analysis of medication reconciliation — 1. The MR at entry is performed by the pharmaceutical team as soon as possible after admission. The sequences of the medical conciliation are attributed to the health professionals according to the recommendations of the French National Authority for Health (HAS).
  2. The MR at the discharge is carried out in collaboration between the pharmaceutical and medical teams. It associates the patient through pharmaceutical interview and relies on the sharing of informations related to the patient's medical treatments. These informations are synthesized in an output conciliation sheet transmitted in real time by secure messaging to the attending physician and the dispensing pharmacist. In parallel, the liaison letter and the patient discharge order are generated in order to guarantee a perfect homogeneity between all the documents transmitted at the patient's exit. MR sequences are attributed to health professionals according to the recommendations of the HAS.

SUMMARY:
Among the strategies to secure the patient's care path, medication reconciliation is a powerful approach for the prevention and interception of medication errors.

DETAILED DESCRIPTION:
All medication errors are not serious. Nevertheless 4 studies show that respectively 5.6%, 5.7%, 6.3% and 11.7% of the medication errors intercepted by medication reconciliation (MR) could have had major, critical or catastrophic consequences for patients. If the consequences of a medication error have a clinical or institutional translation for the patient, they can also directly impact the hospital or caregivers, for example by extending the average length of stay or by increasing the number of consultations or readmissions.

The efficiency of the medication reconciliation approach has never been evaluated in France in comparison with standard care. Before initiating cost-effectiveness studies, we propose to conduct a micro-costing study to evaluate the production costs of this conciliation approach.

The costs are almost exclusively related to human resources and the present study will assess the time spent by the different actors involved in the process.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years old
* Patient non-institutionalized at entry
* For MR :

  * Entry : patients admitted at UMIP between 09/04/2017 and 10/31/2017
  * Discharge : patients returning home or going to a rehabilitation service between 04/09/2017 and 31/10/2017 and having received MR evaluation

Exclusion Criteria:

* Patients not returning home
* Refusal of participation
* Major persons subject to legal protection (safeguard of justice, guardianship), persons deprived of their liberty

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 65 years admitted at the UMIP of Rennes University Hospital between 09/04/2017 and 10/31/2017.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Time spent by professionals | At the inclusion day
  Evaluation of the time spent by each professionals involved in the completion of each step of the MR process.
Average cost of MR process | At the inclusion day
  Evaluation of average cost of MR process at UMIP. Only costs related to human resources are considered.
Number of unintentional discrepancies detected | At the inclusion day
  Number of unintentional discrepancies detected during MR at admission of patients at UMIP.
Severity of unintentional discrepancies detected | At the inclusion day
  Severity of unintentional discrepancies detected during MR at admission of patients at UMIP. Evaluation based on the algorithm provided by the HAS.

CONTACTS AND LOCATIONS:
Overall Officials: Berengere CADOR, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: No